CLINICAL TRIAL: NCT00342485
Title: In Vitro Study of Peripheral Blood Mononuclear Cell Function in Healthy Individuals and Patients
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999993010; OH93-NC-N010
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-03

CONDITIONS: Cell Function
Keywords: Cellular Immunity; HIV-infected; Immune Deficiency; Cancer; Transplantation
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Neoplasms

SUMMARY:
Peripheral blood mononuclear cells (PBMC) will be collected from healthy volunteers and patients who present with different diseases that involve or implicate the immune system dysregulation (HIV infection, autoimmune diseases and cancer). These PBMC will be studied in vitro for a number of functional parameters, including generating soluable factors that inhibit HIV infection, developing patterns of immune dysregulation, and inducing apoptotic T cell death. The purpose of such studies is to obtain insight into the mechanisms of natural resistance to viral infections, AIDS pathogenesis, and disease-induced immune dysregulation.

DETAILED DESCRIPTION:
Peripheral blood mononuclear cells (PBMC) will be collected from healthy volunteers and patients who present with different diseases that involve or implicate the immune system dysregulation (HIV infection, autoimmune diseases and cancer). These PBMC will be studied in vitro for a number of functional parameters, including generating soluable factors that inhibit HIV infection, developing patterns of immune dysregulation, and inducing apoptotic T cell death. The purpose of such studies is to obtain insight into the mechanisms of natural resistance to viral infections, AIDS pathogenesis, and disease-induced immune dysregulation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Greater than or equal to 18 years old.

Documented HIV infection by current DoD criteria (1 ELISA, 2 Confirmatory Western Blot) or by one of the following tests; DNA PCR, RNA PCR, p24 antigen test, viral culture assay.

CD4 lymphocyte cell count greater than 300 mm(3).

EXCLUSION CRITERIA:

Unable to provide informed consent.

Unable to meet the minimum (150 days) and maximum (395 days) research visit interval requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000
Dates: Start 1993-04-12; Study Completion 2008-03-03

CONTACTS AND LOCATIONS:
Locations (1):
- Willford Hall USAF Medical Center, San Antonio, Texas, United States